CLINICAL TRIAL: NCT02658253
Title: Phase Ia/Ib, Randomized, Double Blinded, Dose Escalation Trial to Evaluate the Safety and Immunogenicity in Healthy European and Burkinabe Adults of a Placental Malaria Vaccine Candidate (PRIMVAC) Formulated With Alhydrogel ® or GLA-SE
Brief Title: Trial to Evaluate the Safety and Immunogenicity of a Placental Malaria Vaccine Candidate (PRIMVAC ) in Healthy Adults
Acronym: PRIMALVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Vaccine Initiative (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); Centre national de recherche et de formation sur le paludisme (Other Government); EUCLID Clinical Trial Platform (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C14-60; 2015-002246-31 (EudraCT Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-18 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Malaria
Keywords: Placental malaria vaccine; Plasmodium; PRIMALVAC
MeSH Terms: conditions — Malaria | interventions — glucopyranosyl lipid-A; Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Group A1:Primvac 20 µg +alhydrogel (Experimental): Group A1: 3 European volunteers 0.5 ml intramuscular injection: 20 µg Primvac+ 0.85 mg Alhydrogel®
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: Alhydrogel
- Group A2:Primvac 20 µg +GLA-SE (Experimental): Group A2: 3 European volunteers 0.5 ml intramuscular injection:20 µg Primvac+ 2.5 µg GLA-SE Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: GLA-SE
- Group B1:Primvac 50 µg +alhydrogel (Experimental): Group B1: 6 European volunteers 0.5 ml intramuscular injection: 50 µg Primvac+ 0.85 mg Alhydrogel®
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: Alhydrogel
- Group B2:Primvac 50 µg +GLA-SE (Experimental): Group B2: 6 European volunteers 0.5 ml intramuscular injection:50 µg Primvac+ 2.5 µg GLA-SE Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: GLA-SE
- Group C1:Primvac 50 µg +alhydrogel (Experimental): Group C1: 10 African volunteers 0.5 ml intramuscular injection: 50 µg Primvac+ 0.85 mg Alhydrogel®
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: Alhydrogel
- Group C2: Primvac 50 µg +GLA-SE (Experimental): Group C2: 10 African volunteers 0.5 ml intramuscular injection: 50 µg Primvac+ 2.5 µg GLA-SE
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: GLA-SE
- Group C3: Placebo (Placebo Comparator): Group C3: 5 African volunteers 0.5 ml intramuscular injection: NaCl 0.9% (placebo)
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: Placebo
- Group D1:Primvac 100 µg +alhydrogel (Experimental): Group D1: 10 African volunteers 0.6 ml intramuscular injection: 100µg Primvac+ 0.85 mg Alhydrogel®
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: Alhydrogel
- Group D2: Primvac 100 µg +GLA-SE (Experimental): Group D2: 10 African volunteers 0.6 ml intramuscular injection: 100 µg Primvac+ 2.56 µg GLA-SE
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: PRIMVAC; Biological: GLA-SE
- Group D3: placebo (Placebo Comparator): Group D3: 5 African volunteers 0.6 ml intramuscular injection: NaCl 0.9% (placebo)
  Vaccination schedule: D0, D28 and D56
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PRIMVAC — 3 different dosages of VAR2CSA protein (20µg - 50µg and 100µg)
  Arms: Group A1:Primvac 20 µg +alhydrogel; Group A2:Primvac 20 µg +GLA-SE; Group B1:Primvac 50 µg +alhydrogel; Group B2:Primvac 50 µg +GLA-SE; Group C1:Primvac 50 µg +alhydrogel; Group C2: Primvac 50 µg +GLA-SE; Group D1:Primvac 100 µg +alhydrogel; Group D2: Primvac 100 µg +GLA-SE
Biological: GLA-SE — 2.56 µg of GLA content
  Arms: Group A2:Primvac 20 µg +GLA-SE; Group B2:Primvac 50 µg +GLA-SE; Group C2: Primvac 50 µg +GLA-SE; Group D2: Primvac 100 µg +GLA-SE
Biological: Alhydrogel — 0.85 mg og Aluminium content
  Arms: Group A1:Primvac 20 µg +alhydrogel; Group B1:Primvac 50 µg +alhydrogel; Group C1:Primvac 50 µg +alhydrogel; Group D1:Primvac 100 µg +alhydrogel
Biological: Placebo — 0.9% Na cl
  Arms: Group C3: Placebo; Group D3: placebo

SUMMARY:
The primary objective of the study is to evaluate the safety of 3 different dosages (20µg - 50µg and 100µg) of a placental malaria vaccine candidate (PRIMVAC vaccine) adjuvanted either with Alhydrogel® or GLA-SE, and administered at D0, D28 and D56 in healthy European and Burkinabe adults.

The safety and the tolerability of the vaccine will be assessed on the rate of solicited and unsolicited events/reactions The safety profile will included local and systemic reactions/events as well as the biological safety, based on a clinically significant change of the baseline value of the main biological criteria

DETAILED DESCRIPTION:
The project aims are:

* Primary objective is to evaluate the safety of 3 different dosages (20µg - 50µg and 100µg) of the PRIMVAC vaccine adjuvanted either with Alhydrogel® or GLA-SE, and administered at D0, D28 and D56 in healthy European and Burkinabe adults.
* Secondary objectives are to assess:

  * the humoral immune response to the PRIMVAC vaccine antigen (VAR2CSA) by measuring the variation in the level of total IgG and the level of the isotypic subtypes capable of recognizing the native antigen.
  * the cellular immune response by measuring:

    * the number of T cell secreting IL5 and IFNg following an ex-vivo stimulation with the vaccine antigen
    * the B lymphocyte phenotypes isolated from PBMC
* Exploratory objectives are:

  * To explore the quality of the humoral immune response by the measure of the capability of the antibodies specific to the vaccine antigen to:

    * Cross-react with different VAR2CSA variants expressed on the surface of erythrocytes infected by various strains of Plasmodium falciparum,
    * Inhibit interactions between parasitized erythrocytes expressing different VAR2CSA variants and Chondroitin Sulfate A (receptor involved in placental sequestration),
    * Promote opsonic phagocytosis of parasitized erythrocytes with various strains of Plasmodium falciparum expressing different VAR2CSA variants
  * To explore the quality of the cellular immune response induced by the vaccine antigen by the quantitation of a large panel of cytokines in the ELISpot supernatants.

ELIGIBILITY:
Inclusion criteria (FRANCE):

* Written informed consent (must be obtained prior initiation of any study related intervention)
* Female of age ≥18 years to ≤35 years
* Healthy as a result of review of medical history and/or clinical examination at the time of screening and clinical judgment of the investigator
* Available for the duration of the trial (15 months)
* Willingness to use reliable contraceptive methods such as: birth control pills or birth control patches or vaginal ring, diaphragm, IUD (intrauterine device), condom, progestin implant or injection, or surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation) prior to enrollment at V0 and up to 4 weeks after last vaccination (V6)
* Volunteer reachable by phone during the entire study duration
* Individuals affiliated to a social security regimen
* Volunteer registered in the French Health ministry computerized file and authorized to participate in a clinical trial

Exclusion criteria (FRANCE):

* Pregnancy ongoing as determined by a positive blood test or breastfeeding or lactation.
* Intention to become pregnant during the trial
* Volunteers who are not able to understand and to follow all required study procedures for the whole period of the study in the opinion of the investigator.
* Volunteers with history of any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
* Volunteers participating in any clinical trial with another investigational product 28 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
* History of psychiatric condition that may affect participation in the study (i.e. depression, anti-depressant treatment).
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the study data based on investigator's judgment.
* Any history of malaria infection.
* Travel to a malaria endemic region during the study period or within the six months preceding enrolment in the study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of a serious adverse reaction to any vaccine, including Guillain-Barre Syndrome.
* Administration or planned administration of a vaccine or gammaglobulin not foreseen by the clinical trial protocol within 30 days prior to the first immunization and up to 4 weeks after the last immunization.
* Volunteers with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Administration of immunoglobulins and/or any blood products within the three months preceding the inclusion.
* Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 3 months (inhaled and topical steroids are allowed)
* Seropositive for hepatitis B virus surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Seropositive for human immunodeficiency virus (antibodies to HIV 1-2)
* Any other serious chronic illness requiring hospital specialist supervision.
* Any clinically significant abnormal finding on screening biochemistry or hematology blood tests or urinalysis
* Symptoms, physical signs or laboratory values suggestive of systemic disorders, including infectious renal, hepatic, cardiovascular, pulmonary, cutaneous, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the volunteers.
* Volunteer under guardianship or legal incapacitation.

Inclusion criteria (BURKINA FASO):

* Written informed consent (must be obtained prior initiation of any study related intervention)
* Nulligest Female of age ≥18 years to ≤35 years
* Healthy as a result of review of medical history and/or clinical examination at the time of screening and clinical judgment of the investigator
* Available for the duration of the trial (15 months)
* Willingness to use reliable contraceptive methods such as: birth control pills or birth control patches or vaginal ring, diaphragm, IUD (intrauterine device), condom, progestin implant or injection, or surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation) prior to enrollment at V0 and up to 4 weeks after last vaccination (V6)

Exclusion criteria (BURKINA FASO):

* Pregnancy ongoing as determined by a positive urinary test
* Intention to become pregnant during the trial
* Volunteers who are not able to understand and to follow all required study procedures for the whole period of the study in the opinion of the investigator.
* Volunteers with history of any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
* Volunteers participating in any clinical trial with another investigational product 28 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
* History of psychiatric condition that may affect participation in the study (i.e. depression, anti-depressant treatment).
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data, based on investigator's judgment.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of a serious adverse reaction to any vaccine, including Guillain-Barre syndrome.
* Administration or planned administration of a vaccine or gammaglobulin not foreseen by the clinical trial protocol within 30 days prior to the first immunization and up to 4 weeks after the last immunization.
* Volunteers with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Administration of immunoglobulins and/or any blood products within the three months preceding the inclusion.
* Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 3 months (inhaled and topical steroids are allowed).
* Seropositive for hepatitis B virus surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV).
* Seropositive for human immunodeficiency virus (antibodies to HIV 1-2).
* Any other serious chronic illness requiring hospital specialist supervision.
* Any clinically significant abnormal finding on screening biochemistry or hematology blood tests or urinalysis
* Symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, cutaneous, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the volunteers.
* Volunteer under guardianship or legal incapacitation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09-19 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers with treatment-related adverse events as assessed by FDA scale and the INYVAX EC FP7 Brighton Collaboration Foundation | 35 days
  Grade 3 or higher clinical or laboratory ARI and persisting at Grade 3 for > 48 hours between D0 and D35.

SECONDARY OUTCOMES:
Proportion of volunteer with at least one Serious Adverse Event Following Immunization (SAEFI) for the entire duration of the study | 14 months
  clinical and biological SAEFI and SARI (Serious Adverse Reaction following Immunization (SARI) measured at any time during the volunteer follow-up
Proportion of volunteer with at least one of Adverse Event Following Immunization (AEFI) measured until 1 month post-dose 3 | 3 months
  Immediate AEFI (within 1h following vaccination) as well as unrelated, Related or possibly related solicited and unsolicited AEFI
Proportion of volunteer with at least one Adverse Event Following Immunization (AEFI) measured between M3 and the end of the study (only phase Ia) | 11 months
  Immediate AEFI (within 1h following vaccination) as well as unrelated, Related or possibly related solicited and unsolicited AEFI
Variation in humoral immune response to the vaccine antigen assessed by ELISA | 14 months
  The level of total IgG (g/l): between D0 and the post-vaccination time points M1, M1+7D, M2, M2+7D, M3, M6 and M14
Variation in humoral immune response to the vaccine antigen assessed by ELISA | 3 months
  The level (g/l) of the isotypic subtypes (IgG1, IgG2, IgG3, IgG4) between D0 and the post-vaccination time point M3
Cellular immune responses to the vaccine antigen by Elispot | 63 days
  The median number of spots by ELISpot assay, allowing the counting of IL5 and IFNg secreting cells following an ex-vivo stimulation of PBMC with the vaccine antigen at V0, and 7 days post-dose 1 and 3 (D0- D7 and M2+7D)
Cellular immune responses to the vaccine antigen by FACS | 63 days
  CD19, IgD, CD27, CD38, CD24 and CD43 B lymphocytes subpopulations will be isolated from PBMC at D0 and M2+7D. The data will be expressed for each phenotype as the median percentage of subpopulations among total CD19 B lymphocytes

OTHER OUTCOMES:
Quality of the humoral immune responses | 3 months
  Will be assessed by measuring the capability of the specific vaccine antigen plasma IgGs to:
  * Cross-react with different VAR2CSA variants expressed on the surface of erythrocytes parasitized by various strains of Plasmodium falciparum by flow cytometry.
  * Inhibit interactions between parasitized erythrocytes expressing different VAR2CSA variants and Chondroitin Sulfate A in static and flow conditions
  * Promote opsonic phagocytosis of parasitized erythrocytes with various strains of Plasmodium falciparum expressing different VAR2CSA variants, using the THP1 cell line. Ingestion of fluorescently labeled parasitized erythrocytes by THP1 cells will be assessed by flow cytometry.
Quality of the cellular immune response by the Multiplex technology | 63 days
  Will be assessed by measuring the quantitation of a large panel of cytokines in ELISpot supernatants will be performed at D0- D7 and M2+7D. The difference of the cytokines concentrations (expressed as MFI) between the pre-vaccination samples and the samples collected at D7 and M2+7D will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Professor, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Benoit GAMAIN, Dr, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Sodiomon SIRIMA, Dr, Study Chair — Centre national de recherche et de formation sur le paludisme
Locations (2):
- CNRFP, Ouagadougou, Burkina Faso
- CIC 1417, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chene A, Gangnard S, Guadall A, Ginisty H, Leroy O, Havelange N, Viebig NK, Gamain B. Preclinical immunogenicity and safety of the cGMP-grade placental malaria vaccine PRIMVAC. EBioMedicine. 2019 Apr;42:145-156. doi: 10.1016/j.ebiom.2019.03.010. Epub 2019 Mar 15. PMID 30885725
- [Result] Gamain B, Chene A, Viebig NK, Tuikue Ndam N, Nielsen MA. Progress and Insights Toward an Effective Placental Malaria Vaccine. Front Immunol. 2021 Feb 25;12:634508. doi: 10.3389/fimmu.2021.634508. eCollection 2021. PMID 33717176
- [Result] Sirima SB, Richert L, Chene A, Konate AT, Campion C, Dechavanne S, Semblat JP, Benhamouda N, Bahuaud M, Loulergue P, Ouedraogo A, Nebie I, Kabore M, Kargougou D, Barry A, Ouattara SM, Boilet V, Allais F, Roguet G, Havelange N, Lopez-Perez E, Kuppers A, Konate E, Roussillon C, Kante M, Belarbi L, Diarra A, Henry N, Soulama I, Ouedraogo A, Esperou H, Leroy O, Batteux F, Tartour E, Viebig NK, Thiebaut R, Launay O, Gamain B. PRIMVAC vaccine adjuvanted with Alhydrogel or GLA-SE to prevent placental malaria: a first-in-human, randomised, double-blind, placebo-controlled study. Lancet Infect Dis. 2020 May;20(5):585-597. doi: 10.1016/S1473-3099(19)30739-X. Epub 2020 Feb 4. PMID 32032566